CLINICAL TRIAL: NCT01117714
Title: A Prospective Multicenter Study Comparing Endobronchial and Endoscopic Ultrasound-Guided FNA to Mediastinoscopy/Thoracoscopy in the Staging and Early Detection of Metastases in Lung Cancer
Brief Title: Surgical Versus Non-surgical Staging of Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual was poor at two other sites and manuscript was published which describing another study which accomplished the goals of this project.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A-13245.8; DOD; DOD (Other: Department of Defense)
Record Dates: First submitted 2010-03-25; First posted 2010-05-05 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Lung neoplasm; Pulmonary cancer; Pulmonary neoplasm; Lung cancer staging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS/EBUS with FNA (Active Comparator): EUS/EBUS staging will be performed to evaluate for the presence of mediastinal adenopathy. Each lymph node will be characterized according to published criteria. Staging will follow the TNM system of the AJCC. If present and accessible, at least one lymph node from each accessible station will be aspirated with a separate fine needle using routine FNA and cytological techniques. If multiple lymph nodes are present in a single station, the largest lymph node from that location will be sampled. Patients with cytologically proven mediastinal lymph node metastases (N2 or 3), or those with mediastinal invasion of tumor (T4), will be treated according to standard clinical practice (typically chemotherapy and/or radiotherapy). All complications, morbidity, length of stay attributed to the staging procedures will be recorded at 30 days, or at the time of surgery, whichever is first. All patients will will subsequently undergo surgical resection and complete mediastinal lymph node dissection.
  Interventions: Procedure: Integrated Staging for Early Detection of Metastases in Lung Cancer
- Surgical Mediastinoscopy (Active Comparator): Within two months following CT scan, surgical mediastinoscopy will be performed to evaluate for the presence of mediastinal adenopathy. Each lymph node will be characterized according to published criteria. Staging will follow the TNM system of the AJCC. Patients with cytologically proven mediastinal lymph node metastases (N2 or 3), or those with mediastinal invasion of tumor (T4), will be treated according to standard clinical practice (typically chemotherapy and/or radiotherapy). All complications, morbidity, length of stay attributed to the diagnostic method (medical or surgical) used for staging will be recorded at 30 days, or at the time of surgery, whichever is first. All patients will will subsequently undergo surgical resection and complete mediastinal lymph node dissection.
  Interventions: Procedure: Integrated Staging for Early Detection of Metastases in Lung Cancer

INTERVENTIONS:
Procedure: Integrated Staging for Early Detection of Metastases in Lung Cancer — To determine the accuracy of EBUS/EUS-guided FNA when compared with surgical mediastinoscopy/thoracoscopy

SUMMARY:
About half of all lung cancers are caught after they have spread to nearby lymph nodes. Lymph nodes are small glands found throughout the body that remove bacteria and foreign particles (part of the immune system). A biopsy (tissue sample) can then be sent can be sent to the laboratory for testing. Biopsy results can determine if the cancer has spread (metastases) and to determine the best treatment for a patient with lung cancer.

The purpose of this study is to develop a better way to detect lung cancer earlier before it spreads. This study compares the traditional mediastinoscopy/thoracoscopy surgery with the newer combined Endobronchial Ultrasound (EBUS) and Endoscopic Ultrasound (EUS) -guided fine needle aspiration (FNA) to see if either is better for this purpose. Traditional medical practice is to surgically open the chest and biopsy suspicious lymph nodes (called a mediastinoscopy/thoracoscopy). Some medical centers have already started combining the use of EUS plus EBUS as a standard practice for performing needle biopsy of lymph nodes in the chest to stage and treat lung cancer.

Volunteers for this study have been diagnosed with known or suspected lung cancer, and will receive one of two choices to determine if their cancer has spread:

1. Traditional Surgical Mediastinoscopy/Thoracoscopy Mediastinoscopy is a surgical procedure that allows physicians to view areas of the chest(including the heart, vessels, lymph nodes, trachea, esophagus, and thymus). An endotracheal (within the trachea) tube is inserted followed by a small incision (cut) in the chest. A mediastinoscope is inserted through the incision to see the organs inside the mediastinum and to collect tissue samples. Mediastinoscopy can be used to detect or stage cancer.

   Thoracoscopy is a surgical procedure that involves insertion of a thorascope through a very small incision in the chest wall. A thorascope is a thin, tube-like instrument with a light and lens which usually has a tool for removing tissue. This makes it possible to examine the lungs or other structures in the chest cavity, without making a large incision.
2. EBUS combined with EUS-guided FNA EUS involves the use of a special endoscope fitted with an ultrasound processor at its tip. During EUS, images of surrounding lymph nodes can be obtained and a small needle can be guided through the esophagus into suspicious nodes to biopsy lymph nodes in the chest. Other research studies have shown that using EUS to guide needle biopsy of lymph nodes in the chest is equally if not more accurate than surgical biopsy. However, use of EUS for needle biopsy can limit what is seen by the physician and also limit the sampling of lymph nodes in front of the trachea. EBUS involves the use of a small ultrasound scope that is passed through the opening of the trachea and into the airways. EBUS combined with EUS is a less invasive procedure that provides full view of the lymph nodes in the chest area.

ELIGIBILITY:
Inclusion Criteria:

* Require either surgical or minimally invasive evaluation (EUS/EBUS) of the mediastinum
* Are medically fit to undergo surgery
* Possess known or suspected non-small cell carcinoma of the lung
* Have had PET/CT scan within 45 days of randomization
* Are eligible for complete mediastinal lymph node dissection at surgery if clinically indicated (determined at surgery)

Exclusion Criteria:

* Pathologically documented metastatic disease
* History of malignancy within 5 years other than (skin) basal cell carcinoma
* Bulky mediastinal lymphadenopathy defined as lymph node > 2.0 cm in short axis diameter or contralateral adenopathy or direct invasion mediastinum or great vessels (T4 disease) or have a malignant pleural effusion.
* Peripheral T1 tumors with radiographically normal mediastinum on PET/CT.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of each arm for the staging of lung cancer | Two years
  We will be testing whether or not the sensitivity of the EUS/EBUS technique for identifying malignant mediastinal lymph nodes is more than 10% worse than the sensitivity of the Mediastinoscopy technique. The primary analysis will be a direct comparison of the sensitivities of the 2 measures, where the sensitivity is defined as the number of true positive cases divided by the sum of the true positives and the false negatives, or the proportion of patients who truly have malignant mediastinal lymph nodes that test positive (i.e. via EUS/EBUS or Mediastinoscopy).

SECONDARY OUTCOMES:
Complication rates for each of the diagnostic strategies | At 30 days or at the time of surgery, whichever is first.
  Complication rates associated with each of the diagnostic strategies will be determined based on complications recorded at the time of surgery and up to 30 days after surgery. These complications include morbidity and the length of stay attributed to the diagnostic method.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard A Silvestri, MD, Principal Investigator — Medical University of South Carolina; Brenda J Hoffman, MD, Principal Investigator — Medical University of South Carolina
Locations (3):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina